CLINICAL TRIAL: NCT02361268
Title: End-Stage Renal Disease Intra-dialysis Lifestyle Education Study
Acronym: END-IDLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gurjeet Birdee, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141325; K23AT006965 (NIH)
Record Dates: First submitted 2015-01-29; First posted 2015-02-11 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: End-stage Renal Disease
Keywords: end-stage renal disease; hemodialysis; yoga; mind-body medicine; meditation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-dialysis yoga (Experimental): The experimental intervention in this study is intra-dialysis yoga.
  Interventions: Behavioral: Intradialysis-yoga
- Educational program (Active Comparator): The active comparator for the study is an educational program.
  Interventions: Behavioral: Educational program

INTERVENTIONS:
Behavioral: Intradialysis-yoga — The experimental intervention in this study is intra-dialysis yoga. The intra-dialysis yoga protocol consists of yoga instruction and practice being offered three times a week for 12 weeks. Subjects will have the opportunity to participate in 15 to 60 minutes of yoga during dialysis.
  Arms: Intra-dialysis yoga
Behavioral: Educational program — The educational intervention in this study consists of 12 modules of an educational course, Kidney School, developed and maintained by the Medical Education Institute, Inc. Kidney School is a comprehensive, free, educational curriculum for people with kid
  Arms: Educational program

SUMMARY:
The purpose of this study is to compare the effects of intra-dialysis yoga to an educational program among patients with end-stage renal disease. The investigators hypothesize that yoga as compared to the educational program will significantly improve quality of life.

DETAILED DESCRIPTION:
The investigators propose a prospective, randomized clinical trial among on maintenance hemodialysis to compare the effects of intra-dialysis yoga to an educational program. In a sample of 68 patients the investigators will compare the clinical effects of a 12-week program of yoga to a 12-week education program during dialysis. Outcome assessment of study participants will occur at baseline, 6-weeks, 12-weeks, and 24 weeks for: disease-related quality of life (physical component primary outcome of the study), physical performance, blood pressure, fatigue, satisfaction with dialysis, sleep quality, and mood. Among a sub-sample of 20 participants, the investigators will measure the potential effects of the interventions on endothelial function, arterial stiffness, and autonomic tone. The sub-study will collect outcomes at baseline and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis for ≥3 or months
* Adequately dialyzed (Kt/V ≥1.2 measured within last 3 months)
* Expected to remain in present hemodialysis shift for next 4 months
* Expected to remain on hemodialysis for at least 6 months
* 18 years or older

Exclusion Criteria:

* Acute or chronic medical conditions that would make intra-dialysis yoga potentially hazardous
* Unstable cardiac disease e.g. angina, life threatening arrhythmia
* Chronic lung disease that prevents gentle exercise or deep breathing exercises
* Active cerebrovascular disease
* Major depression
* Chronic symptoms of nausea, vomiting, or diarrhea
* Current participation in exercise or mind body program/practice
* Cognitive impairment (MME ≤ 24) measured at baseline testing visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Physical Component Summary of Kidney Disease Quality of Life-36 questionnaire at 6 weeks, 12 weeks, and 24 weeks. | Baseline, 6 weeks, 12 weeks, and 24 weeks
  The Kidney Disease Quality of Life-36 instrument is a 36-item instrument that contains a generic core (Short Form-12) plus the burden of kidney disease, symptoms/problem of kidney disease, and effects of kidney disease scales.

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Fatigue | Baseline, 6, 12, and 24 weeks
  Questionnaire to assess fatigue among chronic disease patients
Profile of Mood States | Baseline, 6, 12, and 24 weeks
  Questionnaire to assess emotional states
Center for Epidemiological Studies Depression | Baseline, 6, 12, and 24 weeks
  Questionnaire to assess depressive symptoms
End-stage renal disease: Patient satisfaction | Baseline, 6, 12, and 24 weeks
  Questionnaire to assess patient satisfaction with dialysis treatment
Pittsburgh Sleep Quality Index | Baseline, 6, 12, and 24 weeks
  Questionnaire to assess sleep quality
Self-efficacy for self-management | Baseline, 6, 12, and 24 weeks
  Questionnaire to assess self-efficacy for self-management
6-minute walk test | Baseline, 12, and 24 weeks
  Assessment of physical performance
Blood pressure | Baseline and weekly over 12 week study period
Measure of endothelial function with flow-mediated vasodilatation | Baseline and 12-weeks
  Sub-set of patients will have this assessment of endothelial function which measures percentage change in diameter measured in millimeters
Measure of arterial stiffness from radial artery based pulse wave analysis | Baseline and 12-weeks
  Sub-set of patient will have this assessment of arterial stiffness as augmentation index
Autonomic tone | Baseline and 12-weeks
  Assessment of cardiovagal and sympathoneural functioning including baroreflex and heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Gurjeet S Birdee, MD MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553